CLINICAL TRIAL: NCT06968793
Title: Use of Endotracheal Tube Cuff Pressure to Assess Inspiratory Effort During Pressure Support Ventilation: a Prospective Physiological Study
Brief Title: Use of Endotracheal Tube Cuff Pressure to Assess Inspiratory Effort During Pressure Support Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Head of Emergency and Critical Care Center, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIT2025-034-002
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Critical Care; Inspiratory Effort
Keywords: Esophageal pressure; mechanical ventilation; Endotracheal tube cuff pressure; inspiratory effort

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pressure support 15 (Experimental): Pressure support of 15 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 15
- Pressure support 13 (Experimental): Pressure support of 13 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 13
- Pressure support 11 (Experimental): Pressure support of 11 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 11
- Pressure support 9 (Experimental): Pressure support of 9 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 9
- Pressure support 7 (Experimental): Pressure support of 7 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 7
- Pressure support 5 (Experimental): Pressure support of 5 cm H2O will be applied for 5 minutes.
  Interventions: Procedure: Pressure support 5

INTERVENTIONS:
Procedure: Pressure support 15 — Pressure support of 15 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 15
Procedure: Pressure support 13 — Pressure support of 13 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 13
Procedure: Pressure support 11 — Pressure support of 11 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 11
Procedure: Pressure support 9 — Pressure support of 9 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 9
Procedure: Pressure support 7 — Pressure support of 7 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 7
Procedure: Pressure support 5 — Pressure support of 5 cm H2O will be applied for 5 minutes.
  Arms: Pressure support 5

SUMMARY:
During pressure support ventilation (PSV), monitoring of Esophageal Pressure (Pes) has long been considered the gold standard for assessing intrathoracic pressure and the state of respiratory mechanics.The aim of this study was to investigate the correlation between Cuff Pressure (Pcuff) and Esophageal Pressure in patients undergoing tracheal intubation or tracheotomy, and to assess whether Pcuff can be used as a surrogate for Pes for reflecting changes in intrathoracic pressure.The correlation and its consistency between the two under different ventilation conditions were analysed by synchronously monitoring the ΔPcuff and ΔPes to further validate the potential application value of cuff pressure in clinical practice.The results of the study will provide a more convenient and non-invasive method of monitoring intrathoracic pressure in mechanically ventilated patients, thus optimising ventilation strategies, reducing complications, and promoting the innovation and development of monitoring technology in the field of critical care medicine.

DETAILED DESCRIPTION:
Monitoring of Esophageal pressure (Pes) has long been regarded as the gold standard for assessing intrathoracic pressure and respiratory mechanics. The measurement of Esophageal pressure provides indirect information about pleural pressure, which is critical for understanding respiratory mechanics, optimizing mechanical ventilation strategies, and evaluating respiratory muscle load.

However, despite its clinical significance, Esophageal pressure monitoring involves a relatively complex and invasive procedure. Measurement typically requires the insertion of an esophageal catheter via the nasopharyngeal or oropharyngeal route, which may cause patient discomfort and prove challenging in certain cases (e.g., esophageal pathologies or anatomical abnormalities). Consequently, while esophageal pressure remains the current gold standard for evaluating intrathoracic pressure, its clinical application faces limitations.

In contrast, Cuff pressure (Pcuff) monitoring in intubated or tracheostomized patients is simpler and routinely performed. Cuff pressure measurement primarily ensures tracheal tube sealing to prevent gas leakage and aspiration, while also reducing the risk of ventilator-associated pneumonia (VAP). Our preliminary exploratory studies have revealed correlations between Cuff pressure fluctuations and Esophageal pressure, particularly in patients undergoing pressure support ventilation. This finding suggests the potential utility of Cuff pressure as a surrogate marker for intrathoracic pressure. Esophageal pressure inherently reflects pleural pressure through Esophageal pressure changes, while the artificial airway cuff-positioned above the carina within the trachea-detects subtle pressure variations induced by adjacent muscle activity during forceful breathing. These measurements may indirectly indicate inspiratory effort. Variations in cuff positioning might influence results, and our exploratory attempts demonstrated strong waveform correlations between Cuff pressure and Esophageal pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated patients who can tolerate pressure support ventilation (PSV) mode;
2. Respiratory stability: Ability to breathe spontaneously and effectively clear secretions via coughing; oxygen saturation (SpO₂) >90% or a partial pressure of oxygen (PaO₂)/FiO₂ ratio ≥150 mmHg when the ventilator's oxygen concentration is set to 40%;
3. Hemodynamic stability: Heart rate (HR) ≤120 bpm, systolic blood pressure (SBP) 90-150 mmHg, with no vasoactive agents or norepinephrine dosage ≤0.1-0.2 μg/kg·min (or equivalent doses of other vasoactive agents);
4. Metabolic stability, with an esophageal pressure monitoring catheter already placed prior to the trial;
5. Written informed consent obtained from the patient or their legal guardian.

Exclusion Criteria:

1. Age <18 years;
2. Pregnancy;
3. Hemodynamic instability: Mean arterial pressure (MAP) <60 mmHg, heart rate (HR) >120 bpm or <60 bpm;
4. Respiratory instability: Respiratory rate (RR) >35 bpm or oxygen saturation (SpO₂) <90%;
5. Neuromuscular disorders or phrenic nerve injury;
6. Recent trauma or surgery involving the trachea, esophagus, neck, or thorax, contraindications to esophageal catheter insertion, or inability to monitor esophageal pressure;
7. High bleeding risk: Severe coagulopathy/bleeding disorders, esophageal/gastric varices, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Tidal swing of endotracheal tube cuff pressure (ΔPcuff) | From enrollment to the end of treatment at 4 hours
  Tidal swing of endotracheal tube cuff pressure (ΔPcuff) will be measured.
Tidal swing of esophageal pressure (∆Pes) | From enrollment to the end of treatment at 4 hours
  Tidal swing of esophageal pressure (∆Pes) will be measured.
Esophageal pressure-time product (PTP) | From enrollment to the end of treatment at 4 hours
  Esophageal pressure-time product (PTP) will be measured.
Inspiratory muscle pressure (Pmus) | From enrollment to the end of treatment at 4 hours
  Inspiratory muscle pressure (Pmus) will be measured.

SECONDARY OUTCOMES:
Occluded airway pressure at 100ms (P0.1) | From enrollment to the end of treatment at 4 hours
  Occluded airway pressure at 100ms (P0.1) will be measured.
Maximal decrease of airway pressure during end-expiratory occlusion (∆Pocc) | From enrollment to the end of treatment at 4 hours
  Maximal decrease of airway pressure during end-expiratory occlusion (∆Pocc) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No